CLINICAL TRIAL: NCT01293994
Title: A Study of Genetic Variation Influencing Pain and Response to Opioid Medications in Patients With Chronic Pain
Brief Title: A Study of Genetic Variation Influencing Pain and Response to Opioid Medications
Status: Withdrawn | Type: Observational
Why Stopped: Do not have necessary resources to continue
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Larry Fu-nien Chu, Professor of Anesthesia, Stanford University
Other Study IDs: SU-11222010-7229; IRB #16198 (Other: Stanford University Panel on Human Subjects)
Record Dates: First submitted 2011-02-09; First posted 2011-02-11 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Pain
Keywords: Chronic Pain, Genetic Variation, Opioid Medications, Pain
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva biospecimen collection will be performed via mail or in person. The PI will send participants a letter informing them of the opportunity to participate in a study of genetic variation influencing pain and opioid responsiveness phenotypes. If participants agree to provide a saliva biospecimen and to participate in the study, an informed consent letter and an Oragene™ DNA Self-Collection Kit, in disk format OG-250 (DNA Genotek, Inc., Ottawa, Ontario, Canada) will be sent to the participant by the PI. According to the manufacturer instructions, participants will provide a 2 ml saliva sample, which will be preserved using the reagents provided within the Oragene™ kit. Saliva samples are considered stable at room temperature for 5 years by Oragene™.
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will be collecting saliva DNA samples from chronic back pain patients. The investigators hope to find candidate genes associated with response to opioid medication by correlating molecular genetics data with pain measurement and opioid responsiveness data including opioid hyperalgesia and opioid analgesic tolerance.

DETAILED DESCRIPTION:
The investigators hope to find a genetic association with various physiologic responses to opioid medication in patients who suffer from chronic pain (e.g. OIH vs. analgesic tolerance, baseline pain sensitivity, etc.). This has never been done before, and if it proves successful, it could provide physicians a greater understanding of why some chronic opioid users continue needing increased doses of opioids. This data may also help predict which patients will do well with chronic opioid therapy and which ones may not. Initial data with OPRM1 gene analysis in humans already implicates certain SNPs with opioid responsiveness and there have been suggestions for screening patients for OPRM1 prior to initiating opioid therapy in order to optimize their treatment response (Reynolds et al., 2008).

Clin Lab Med. 2008 Dec;28(4):581-98. The value of CYP2D6 and OPRM1 pharmacogenetic testing for opioid therapy. Reynolds KK, Ramey-Hartung B, Jortani SA.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient, aged 18-71
2. Recipient of chronic opioid therapy
3. Patient is able to produce a saliva sample
4. If a past study participant, patient will have agreed to be contacted for future studies.

Exclusion Criteria:

a. not meeting inclusion criteria

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any gender, ages 18-70, of any ethnic background
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Genetic association with various physiologic responses to opioid medication in patients | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Larry Fu-nien Chu, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No